CLINICAL TRIAL: NCT05397899
Title: Effects of Abdominal Hypopressive Technique on Postpartum Low Back Pain
Brief Title: Abdominal Hypopressive Technique on Postpartum Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Asma Bhatti
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Postpartum

STUDY DESIGN:
Intervention Model Description: This will be a Pretest-Postest Control group Design with parallel assignment of patients into two groups.
Who Masked: Outcomes Assessor
Masking Description: outcome assessor will be kept blind about the group of patients and treatment received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AHT group (Experimental): This group will receive Abdominal hypopressive exercises. Each AHT will be repeated 3-5 times with 1 min rest between exercises (shift to new posture, lying,sitting and standing). Between 6 and 15 hypopressive exercises (HEs) will be performed within each session based on the participant's mastery of the exercises and readiness to progress, for 6 weeks.
  Interventions: Other: Abdominal hypopressive Exercises (AHE)
- General exercise group (Active Comparator): This group will receive general exercises (Bridging, knee to chest, Straight leg rise) these will be repeated 3-5 times with 1 min rest between exercises. Between 6 and 15 repetitions will be performed within each session based on the participant's mastery of the exercises and readiness to progress. Each exercise to be repeated 3-5 times per set, and participants will be asked to perform technique once daily for 6 weeks
  Interventions: Other: General exercises

INTERVENTIONS:
Other: Abdominal hypopressive Exercises (AHE) — Active and specific Therapeutic exercises will be used to treat postpartum low back pain in this study. AHE consisted of exhaling to their expiratory reserve volume, then holding their breath (apnea), and expanding their rib cage, to draw their abdominal wall inward and cranially without inhalation. Each exercise will have a specific frequency, intensity, and duration.
  Arms: AHT group
Other: General exercises — General exercises are therapeutic exercises for core muscles for the treatment of postpartum low back pain.
  Arms: General exercise group

SUMMARY:
Postpartum Low back pain (PP-LBP) is more common and can lead to limitations to women's daily activity. Pregnancy related low back pain has been reported to occur in 55% to 78% women worldwide.This study is planned to determine the effects of abdominal hypopressive technique on postpartum low back pain, mobility and disability.

DETAILED DESCRIPTION:
literature suggests the use of hypopressive abdominal techniques to be effective in increasing the thickness of the abdominal muscles and hence add to the stability of the spine and alleviation of low back pain in the postpartum period. This will be a randomized controlled trial, with two groups.

Participants in the experimental group will learn how to perform the "hypopressive maneuver", which consisted of exhaling to their expiratory reserve volume, then holding their breath (apnea), and expanding their rib cage, to draw their abdominal wall inward and cranially without inhalation. control group will perform general exercises. Both groups will be assessed at pre and post test (after 6weeks)

ELIGIBILITY:
Inclusion Criteria:

* Postpartum non-radiating low back Pain
* LBP severity >3 on numeric pain rating scale (NPRS)
* Spontaneous vaginal delivery

Exclusion Criteria:

* Prenatal history of low back pain
* Caesarean section
* Hypertension
* Puerperium period
* Arterial complications
* Neurological deficit
* Disc Bulge
* Lumbar Radiculopathy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Changes from Baseline to 6th week
  The pain score was assessed using the numeric pain rating scale (NPRS) is a scoring system, wherein the pain level was quantified on a scale of 0 (no pain) to 10 (worst possible pain). The NPRS is a valid and frequently employed method of musculoskeletal pain assessment.
Pregnancy Mobility Index | Changes from Baseline to 6th week
  It is self-report mobility scale designed specifically for the pregnant women. The internal consistency (Cronbach's alpha) is 0.8 or higher indicating a good construct validity. The assumptions that the Pregnancy Mobility Index scores increase during pregnancy and decrease after delivery and that women with back or pelvic problems scored higher on the Pregnancy Mobility Index domains than women without back or pelvic pain were confirmed, indicating a good criterion validation.
  Its scores range from 0 to 100, in which 0 equals 'normal performance' and 100 indicates 'maximum disability
Maternal Postpartum Quality of Life Index | Changes from Baseline to 6th week
  It is a sixteen-item scale, which is a valid and reliable instrument for postpartum QOL assessment. It includes items on the different aspects of postpartum QOL and can be used for the early diagnosis of impaired postpartum QOL. The QoL score ranges from 0 to 30, with higher scores indicating higher QoL.

SECONDARY OUTCOMES:
Oswestry Low Back Pain Disability Index(ODI) | Changes from Baseline to 6th week
  The Oswestry Low Back Pain Disability Index is a validated, 10-point patient-reported outcome questionnaire. It is considered the 'gold standard for measuring disability and quality of life (QoL) impairment for adults with low back pain. The Cronbach-α for the ODI is 0.75. The ODI showed excellent test- retest reliability (intraclass correlation coefficient = 0.91)

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Holy Family Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellido-Fernandez L, Jimenez-Rejano JJ, Chillon-Martinez R, Gomez-Benitez MA, De-La-Casa-Almeida M, Rebollo-Salas M. Effectiveness of Massage Therapy and Abdominal Hypopressive Gymnastics in Nonspecific Chronic Low Back Pain: A Randomized Controlled Pilot Study. Evid Based Complement Alternat Med. 2018 Feb 22;2018:3684194. doi: 10.1155/2018/3684194. eCollection 2018. PMID 29681973
- [Background] Saleh MSM, Botla AMM, Elbehary NAM. Effect of core stability exercises on postpartum lumbopelvic pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2019;32(2):205-213. doi: 10.3233/BMR-181259. PMID 30282349
- [Background] Davenport MH, Marchand AA, Mottola MF, Poitras VJ, Gray CE, Jaramillo Garcia A, Barrowman N, Sobierajski F, James M, Meah VL, Skow RJ, Riske L, Nuspl M, Nagpal TS, Courbalay A, Slater LG, Adamo KB, Davies GA, Barakat R, Ruchat SM. Exercise for the prevention and treatment of low back, pelvic girdle and lumbopelvic pain during pregnancy: a systematic review and meta-analysis. Br J Sports Med. 2019 Jan;53(2):90-98. doi: 10.1136/bjsports-2018-099400. Epub 2018 Oct 18. PMID 30337344
- [Background] Da Cuna-Carrera I, Alonso-Calvete A, Soto-Gonzalez M, Lantaron-Caeiro EM. How Do the Abdominal Muscles Change during Hypopressive Exercise? Medicina (Kaunas). 2021 Jul 9;57(7):702. doi: 10.3390/medicina57070702. PMID 34356983
- [Background] Juez L, Nunez-Cordoba JM, Couso N, Auba M, Alcazar JL, Minguez JA. Hypopressive technique versus pelvic floor muscle training for postpartum pelvic floor rehabilitation: A prospective cohort study. Neurourol Urodyn. 2019 Sep;38(7):1924-1931. doi: 10.1002/nau.24094. Epub 2019 Jul 11. PMID 31297874
- [Background] Soriano L, Gonzalez-Millan C, Alvarez Saez MM, Curbelo R, Carmona L. Effect of an abdominal hypopressive technique programme on pelvic floor muscle tone and urinary incontinence in women: a randomised crossover trial. Physiotherapy. 2020 Sep;108:37-44. doi: 10.1016/j.physio.2020.02.004. Epub 2020 Feb 19. PMID 32707289